CLINICAL TRIAL: NCT00352001
Title: A Phase I/II Study of Revlimid (Lenalidomide) in Combination With Vidaza (Azacitidine) in Patients With Advanced Myelodysplastic Syndrome (MDS)
Brief Title: Lenalidomide and Azacitidine in Treating Patients With Advanced Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mikkael Sekeres MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mikkael Sekeres MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE17Z05; P30CA016042 (NIH); UCLA-0511032-01; UCLA-RDN-5405; UCLA-05011032-01; CASE17Z05 (Other: Case Comprehensive Cancer Center); NCT00326846 (obsolete NCT alias)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts; previously treated myelodysplastic syndromes; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and Azacitidine (Experimental)
  Interventions: Drug: azacitidine; Drug: lenalidomide

INTERVENTIONS:
Drug: azacitidine — Azacitidine subcutaneously once daily on days 1-5 or days 1-5 and 8-12. Treatment repeats every 28 days for up to 7 courses in the absence of relapse (after achieving complete or partial remission), disease progression, or unacceptable toxicity.
  Other Names: Vidaza®
Drug: lenalidomide — Oral lenalidomide once daily on days 1-14 or days 1-21.Treatment repeats every 28 days for up to 7 courses in the absence of relapse (after achieving complete or partial remission), disease progression, or unacceptable toxicity.
  Other Names: Revlimid®

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Lenalidomide may also stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Azacitidine may also cause cancer cells to look more like normal cells, and to grow and spread more slowly. Giving lenalidomide together with azacitidine may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lenalidomide and azacitidine in treating patients with advanced myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of lenalidomide and azacitidine in patients with advanced myelodysplastic syndromes (MDS).

Secondary

* Review clinical outcomes, as defined by the International Working Group criteria, in patients treated with this regimen.
* Determine time to transformation to acute myeloid leukemia or death in patients treated with this regimen.
* Determine time to relapse after achieving complete or partial remission in patients treated with this regimen.
* Determine time to disease progression in patients treated with this regimen.
* Determine the effect of this regimen on hematologic status (including peripheral blood counts and the need for platelet and/or red blood cell transfusions) in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study.

Patients receive oral lenalidomide once daily on days 1-14 or days 1-21 and azacitidine subcutaneously once daily on days 1-5 or days 1-5 and 8-12. Treatment repeats every 28 days for up to 7 courses in the absence of relapse (after achieving complete or partial remission), disease progression, or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses and/or increasing dosing frequencies of lenalidomide and azacitidine until the maximum tolerated dose (MTD) is determined or the sixth dose level is reached, whichever occurs first. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first course of therapy.

After completion of study treatment, patients are followed annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS) meeting one of the following criteria:

  * French-American-British histological classification criteria

    * Refractory anemia with excess blasts (RAEB), defined as 5-19% myeloblasts in the bone marrow

      * Patients with 20% blasts are considered to have acute myeloid leukemia (per WHO classification system) and are therefore excluded in this study
    * Chronic myelomonocytic leukemia (CMML), defined as 10-19% myeloblasts in the bone marrow and/or 5-19% blasts in the blood
  * WHO histological classification criteria

    * RAEB-1, defined as 5-9% myeloblasts in the bone marrow
    * RAEB-2, defined as 10-19% myeloblasts in the bone marrow and/or 5-19% blasts in the blood
    * CMML-2, defined as 10-19% myeloblasts in the bone marrow and/or 5-19% blasts in the blood
  * International Prognostic Scoring System (IPSS) score of intermediate 2 (1.5-2.0 points based on karyotype, cytopenias, and bone marrow blast percentage) or high (≥ 2.5 points), in the setting of ≥ 5% myeloblasts
* Considered ineligible for bone marrow transplantation as first-line therapy

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception for 4 weeks before, during, and for 4 weeks after completion of study treatment
* No serious medical condition, laboratory abnormality, or psychiatric illness that, in the opinion of the treating physician, would preclude study participation or preclude giving informed consent
* No preexisting neurotoxicity or neuropathy ≥ grade 2
* No rash or prior hypersensitivity or allergic reaction ≥ grade 3 to thalidomide
* Creatinine ≤ 2.0 mg/dL
* AST and ALT ≤ 2.0 times upper limit of normal
* Bilirubin ≤ 2 mg/dL
* Platelet count ≥ 50,000/mm^3
* Absolute neutrophil count ≥ 500/mm^3
* No other malignancy within the past 3 years except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No history of thromboembolic event or other condition requiring use of anticoagulation with warfarin or low molecular-weight heparin
* No known or suspected hypersensitivity to azacitidine or mannitol

PRIOR CONCURRENT THERAPY:

* More than 28 days since prior and no other concurrent investigational agents for MDS
* More than 28 days since prior approved therapy for MDS
* More than 14 days since prior growth factors
* More than 28 days since prior and no concurrent supraphysiologic doses (equivalent to > 10 mg/day of prednisone) of corticosteroids
* More than 12 months since prior radiotherapy, chemotherapy, or cytotoxic therapy for treatment of conditions other than MDS
* No prior lenalidomide or azacitidine
* No prior stem cell or bone marrow transplantation
* No concurrent androgens, epoetin alfa, or chemotherapy for MDS

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael A. Sekeres, MD, MS, Study Chair — The Cleveland Clinic
Locations (3):
- United States (3):
  - University of California at Los Angeles, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Cleveland Clinic Taussig Cancer Instititute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Sekeres MA, Tiu RV, Komrokji R, Lancet J, Advani AS, Afable M, Englehaupt R, Juersivich J, Cuthbertson D, Paleveda J, Tabarroki A, Visconte V, Makishima H, Jerez A, Paquette R, List AF, Maciejewski JP. Phase 2 study of the lenalidomide and azacitidine combination in patients with higher-risk myelodysplastic syndromes. Blood. 2012 Dec 13;120(25):4945-51. doi: 10.1182/blood-2012-06-434639. Epub 2012 Aug 22. PMID 22915641

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide and Azacitidine
Started | 37
Azacitidine 75mg/Lenalidomide 5mg-14 Day | 3
Azacitidine 75mg/Lenalidomide 5mg-21 Day | 3
Azacitidine 75mg/Lenalidomide 10mg-14day | 3
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 76.5 [54 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: PHASE I: Maximum Tolerated Dose of Azacitidine
Description: Participants will be enrolled on the Phase I study portion in blocks of 3 to varying doses of Revlimid® (lenalidomide) and Vidaza® (azacitidine) (Table 1). To determine the MTD, a standard "3+3" design will be used. DLT will be assessed during the first cycle of therapy within each treatment group. No Maximum dose was reach but the go-forward dose agreed upon by the investigators is reported here.
Time Frame: After 1 courses (1 months)
Population: Participants in Phase I
Measure: Number; unit: mg/m2 subcutaneously for 5 days
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 18
mg/m2 subcutaneously for 5 days | 75

2. Primary Outcome: PHASE II: Determine the Number of Patients With Responses for Efficacy(Measured as Response Rate)
Description: For the Phase II study portion, to determine the efficacy (measured as response rate) of the combination therapy as defined by the International Working Group (IWG) criteria (CR, complete remission; PR, partial remission; or HI, hematological improvement.
  Complete response (CR) is defined as: Disappearance of the chromosomal abnormality without appearance of new ones.
  Partial response (PR) is defined as: At least 50% reduction of the chromosomal abnormality.
  Hematologic Improvement (HI) is defined as: red blood cell increase of >=1.5g/dL, a platelet response of >=30X10^9/L or by at least 100% for values starting <20X10^9/L, or a neutrophil response of at least 100% and absolute increase of >0.5X10^9/L
Time Frame: After 4 courses (4 months)
Population: Intention to Treat
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 37
participants | 26

3. Primary Outcome: PHASE II: Determine the Number of Patients With Responses for Efficacy(Measured as Response Rate)
Description: For the Phase II study portion, to determine the efficacy (measured as response rate) of the combination therapy as defined by the International Working Group (IWG) criteria (CR, complete remission; PR, partial remission; or HI, hematological improvement)
  Complete response (CR) is defined as: Disappearance of the chromosomal abnormality without appearance of new ones.
  Partial response (PR) is defined as: At least 50% reduction of the chromosomal abnormality.
  Hematologic Improvement (HI) is defined as: red blood cell increase of >=1.5g/dL, a platelet response of >=30X10^9/L or by at least 100% for values starting <20X10^9/L, or a neutrophil response of at least 100% and absolute increase of >0.5X10^9/L
Time Frame: After 7 courses (months)
Population: Intention to Treat
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 37
participants | 26

4. Secondary Outcome: Time to Transformation to Acute Myeloid Leukemia or Death
Description: Time (in months) patients took to evolve to myeloid leukemia or death after achieving a complete response using the RECIST criteria
Time Frame: After 7 months of treatment, until the date of first documented myeloid leukemia or death, whichever came first, assessed up to 55 months
Population: Patients who achieved a complete response
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 16
months | 13.6 [3 to 55]

5. Secondary Outcome: Time to Relapse After Achieving Complete Response
Time Frame: as for outcome 4
Population: Only patients with a complete response were analysed
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 16
months | 17 [3 to 39]

6. Secondary Outcome: Number of Patients That Experience Grade 3 or 4 Treatment Related Non-hematologic Adverse Events
Time Frame: After 7 months
Population: Intention to Treat
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 37
participants | 9

7. Primary Outcome: PHASE I: Maximum Tolerated Dose of Lenalidomide
Description: as for outcome 1
Time Frame: After 1 courses (1 months)
Population: Participants in Phase I
Measure: Number; unit: mg orally for 21 days
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 18
mg orally for 21 days | 10

8. Secondary Outcome: Overall Survival Among Patients With Complete Response
Description: Time (in months) patients who achieved a complete response using the RECIST criteria were alive on study
Time Frame: as for outcome 4
Population: Only patients with complete response
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Azacitidine
Number analyzed (Participants) | 16
months | 37 [7 to 55]

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Lenalidomide and Azacitidine
Serious Adverse Events (participants affected / at risk) | 10/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Azacitidine (N=37)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (6)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
CNS Hemorrhage/bleeding (Nervous system disorders) | 1 (1)
Deep vein or cardiac thrombosis (Vascular disorders) | 1 (1)
general disorder (General disorders) | 1 (1)
weakness/dizziness (Nervous system disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Hemoglobin for leukemia studies (Investigations) | 1 (1)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Increased blood urea nitrogen (BUN) (Investigations) | 1 (1)
Neutrophils/granulocytes (Investigations) | 2 (4)
Platelets (Investigations) | 2 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — Catheter Related Infection
Constitutional Symptom (General disorders) | 1 (1) — Sudden death on study - unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Azacitidine (N=37)
Cardiac Arrhythmia - Other (Cardiac disorders) | 3 (3)
Cardiac General - Other (Cardiac disorders) | 3 (4)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 3 (4)
Infection with unknown ANC (Infections and infestations) | 3 (3)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 3 (3)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 4 (4)
Weight loss (Investigations) | 4 (4)
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (4)
Taste alteration (dysgeusia) (Nervous system disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (5)
Hemorrhage/Bleeding - Other (Vascular disorders) | 4 (7)
Rigors/chills (General disorders) | 5 (5)
Gastrointestinal - Other (Gastrointestinal disorders) | 5 (9)
Edema: limb (General disorders) | 5 (5)
Neurology - Other (Psychiatric disorders) | 5 (7)
Hypotension (Vascular disorders) | 6 (8)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 6 (6)
Infection - Other (Infections and infestations) | 6 (8)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Constitutional Symptoms - Other (General disorders) | 8 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 10 (11)
Dizziness (Nervous system disorders) | 10 (10)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 11 (19)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 11 (14)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Leukocytes (total WBC) (Investigations) | 12 (34)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 12 (17)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (19)
Hemoglobin (Blood and lymphatic system disorders) | 16 (29)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 17 (29)
Injection site reaction/extravasation changes (General disorders) | 17 (20)
Platelets (Investigations) | 18 (43)
Diarrhea (Gastrointestinal disorders) | 18 (24)
Pain (General disorders) | 19 (36)
Constipation (Gastrointestinal disorders) | 20 (22)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes